CLINICAL TRIAL: NCT05070429
Title: Randomized Trial of Telehealth vs. Conventional Hearing Care Delivery in the ACHIEVE Study
Brief Title: ACHIEVE Hearing Intervention Follow-Up Study
Acronym: ACHIEVE-HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of North Carolina (Other); University of South Florida (Other); University of Minnesota (Other); University of Mississippi Medical Center (Other); Wake Forest University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00284937; R01DC019408 (NIH)
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss; Aging
Keywords: hearing healthcare; telehealth hearing healthcare; clinic-based hearing healthcare; hearing healthcare service delivery models
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional hearing healthcare group (Other): The conventional hearing healthcare group will have clinic-based visits every 6 months for the duration of the 2-year study. During Year 1, this group will receive clinic-based audiological rehabilitative service delivery and be able to use conventional options to address any unanticipated needs that arise, and then during Year 2, this group will also receive telehealth audiological rehabilitative service delivery and be able to utilize telehealth options, in addition to conventional options, to address any unanticipated needs that arise.
  Interventions: Other: Clinic-based audiological rehabilitative service delivery; Other: Telehealth audiological rehabilitative service delivery
- Telehealth hearing healthcare group (Other): The telehealth hearing healthcare group will have clinic-based visits every 6 months for the duration of the 2-year study. This group will receive telehealth audiological rehabilitative service delivery and be able to utilize telehealth options, in addition to conventional options, to address any unanticipated needs that arise during both years of the study.
  Interventions: Other: Telehealth audiological rehabilitative service delivery

INTERVENTIONS:
Other: Clinic-based audiological rehabilitative service delivery — Participants will have scheduled clinic-based visits at 6 and 12 months post-randomization to reinforce self-management strategies and perform hearing aid checks.
  Other Names: Conventional hearing healthcare
  Arms: Conventional hearing healthcare group
Other: Telehealth audiological rehabilitative service delivery — Participants' scheduled clinic-based visits will be complemented with asynchronous and synchronous telehealth that will allow for routine troubleshooting of communication challenges, hearing aid technical issues, and reinforcement of self-management support strategies. At an initial session, participants will be instructed in the use of a study-provided, internet-enabled tablet device for telehealth sessions, re-introduced to the hearing loss toolkit for self-management and C2Hear Reusable Learning Objects within the context of the telehealth platform, re-evaluated on the Client Oriented Scale of Improvement (COSI) goals. Two remote follow-up sessions will be scheduled 3 and 6 weeks later to confirm participants' comfort with the telehealth platform and then completed every 6 months, in addition to scheduled 6-month clinic-based visits.
  Other Names: Telehealth hearing healthcare

SUMMARY:
The ACHIEVE Hearing Intervention Follow-Up study is a randomized trial of a telehealth versus conventional clinic-based hearing healthcare (HHC) delivery model among older adults who are existing hearing aid users to determine if a telehealth HHC model improves hearing aid use and other communication outcomes compared to clinic-based HHC.

DETAILED DESCRIPTION:
This study is a multi-site randomized efficacy trial of a telehealth versus conventional clinic-based hearing healthcare (HHC) delivery model among older adults who are existing hearing aid users to determine if a telehealth HHC model improves hearing aid use and other communication outcomes compared to clinic-based HHC.

Participants will be recruited from the ongoing Aging & Cognitive Health Evaluation in Elders (ACHIEVE) randomized trial in which the investigators recruited 977 adults ages 70-84 with untreated mild-to-moderate hearing loss from January 2018 to October 2019 who were randomized to a hearing intervention (i.e., conventional clinic-based delivery of hearing services and technologies) versus a successful aging education control intervention (i.e., one-on-one sessions with a health educator on topics important for healthy aging). From 2021-2022, as participants in the hearing intervention group (fixed sample, n=490) complete the pre-specified three years of follow-up in the ACHIEVE trial, the investigators will recruit these existing hearing aid users and randomize the participants 1:1 to receive continued conventional clinic-based delivery of hearing care services versus a model that incorporates telehealth. Accounting for loss to follow-up and death, the investigators conservatively estimate that n=400 participants currently in the hearing intervention group will be recruited into this two-year follow-up study.

The main analyses will be conducted at one-year post-randomization when hours of hearing aid use (primary outcome) and patient-centered hearing and communication, social functioning, and quality of life secondary outcomes will be contrasted between the two intervention groups.

After one year of follow-up, participants randomized to the conventional HHC arm will cross-over and also receive telehealth HHC, while participants randomized to the telehealth HHC arm will continue to receive telehealth HHC. All participants will continue to be followed for 2 years post-randomization for observational analyses, with data collection follow-up visits occurring every 6 months.

ELIGIBILITY:
To be eligible for the current study, participants must:

* have been eligible for and participated in the hearing intervention arm of the ACHIEVE trial (see original eligibility criteria below)
* agree to be randomized to receive continued hearing care via either a telehealth or conventional delivery model, and
* agree to participate in the follow-up study.

Original ACHIEVE Inclusion Criteria:

* Age 70-84 years
* Community-dwelling, fluent English speaker
* Availability of participant in area for study duration
* Adult-onset hearing impairment, defined as four-frequency pure tone average (PTA, 0.5-4 kilohertz (kHz), better ear) ≥30 decibel (dB) hearing level (HL) (decibels hearing level) & <70 dB HL
* Speech recognition scores in quiet ≥60% in better ear
* Mini-Mental State Exam (MMSE) score ≥23 for participants with high school degree or less, or ≥25 for participants with some college education or more

Original ACHIEVE Exclusion Criteria:

* Reported disability in ≥2 activities of daily living (ADLs)
* Vision impairment (worse than 20/63 on the Minnesota Near Vision Card)
* Self-reported use of a hearing aid in the past 1 year
* Medical contraindication to use of hearing aids (e.g., draining ear)
* Unwilling to wear hearing aids on a daily basis
* Conductive hearing impairment with air-bone gap >15 dB in two or more contiguous frequencies in both ears

Ages: 73 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 339 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2025-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Lin, MD, PhD, Principal Investigator — Johns Hopkins University; Victoria A Sanchez, AuD, PhD, Principal Investigator — University of South Florida
Locations (4):
- United States (4):
  - Johns Hopkins Comstock Center for Public Health Research and Prevention, Hagerstown, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The ACHIEVE data coordinating center, in coordination with the Steering Committee and NIH, will prepare a public access data release that complies with prevailing NIH and HIPAA guidelines in place when the study has been completed. Any participant identifying information will be removed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will share data 1 year following publication of the main results paper for the trial, unless NIH policy dictates that data be shared sooner.
Access Criteria: To be determined

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Hearing Healthcare Group: The conventional hearing group will have clinic-based visits every 6 months for the 2-year study. During Year 1, they will receive clinic-based audiological rehabilitative service and use conventional options to address unanticipated needs. During Year 2, this group will also receive telehealth audiological rehabilitative service delivery and be able to utilize telehealth, and conventional options, to address any unanticipated needs.
  Clinic-based audiological rehabilitative service: Participants will have scheduled clinic-based visits at 6 and 12 months post-randomization to reinforce self-management strategies and hearing aid checks.
  Telehealth audiological rehabilitative service: Participants' scheduled clinic-based visits will be complemented with asynchronous and synchronous telehealth that will allow for routine troubleshooting of communication challenges, hearing aid issues, and reinforcement of self-management support strategies. At an initial session, participants will be instructed in the use of, an internet-enabled tablet device for telehealth sessions, re-introduced to the hearing loss toolkit for self-management and C2Hear Reusable Learning Objects within the context of the telehealth platform, re-evaluated on the Client Oriented Scale of Improvement goals. Two remote follow-up sessions will be scheduled 3 and 6 weeks later to confirm participants' comfort with the telehealth platform, completed every 6 months, and scheduled 6-month clinic-based visits.
Period: Overall Study
Arm/Group | Conventional Hearing Healthcare Group | Telehealth Hearing Healthcare Group
Started | 176 | 163
Completed | 159 | 153
Not Completed | 17 | 10
Not completed — Death | 0 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 15 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Hearing Healthcare Group | Telehealth Hearing Healthcare Group | Total
Number analyzed (Participants) | 176 | 163 | 339
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 176 | 163 | 339
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.7 (3.8) | 79.1 (4.0) | 78.9 (3.9)
Age, Customized [Count of Participants; unit: Participants]
  Age in Categories: Between 72 and 74 years | 27 | 22 | 49
  Age in Categories: 75 - 79 years | 82 | 65 | 147
  Age in Categories: 80 - 84 years | 53 | 56 | 109
  Age in Categories: 85 - 88 years | 14 | 20 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 87 | 186
  Male | 77 | 76 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 170 | 158 | 328
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 18 | 35
  White | 157 | 145 | 302
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 176 | 163 | 339
Site [Count of Participants; unit: Participants]
  Forsyth County, NC | 37 | 35 | 72
  Jackson, MS | 45 | 39 | 84
  Minneapolis, MN | 43 | 42 | 85
  Washington County, MD | 51 | 47 | 98

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Hours of Hearing Aid Use
Description: Average daily hours of hearing aid use is obtained using objective hearing aid data logging. If a participant wears a hearing aid in both ears, then the ear with the greatest number of hours will be selected.
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: Daily hours
Arm/Group | Conventional Hearing Healthcare Group | Telehealth Hearing Healthcare Group
Number analyzed (Participants) | 159 | 153
Daily hours | 7.37 (5.15) | 7.20 (5.05)
Statistical Analysis 1: Comparison: Conventional Hearing Healthcare Group vs Telehealth Hearing Healthcare Group; Used a weighted regression model with an identity link to compare average daily hours of hearing aid use at one-year post-randomization between participants assigned to the telehealth HHC or conventional HHC. Inverse probability of treatment weights will be calculated and included in the model for the primary outcome; Test type: Superiority; p = 0.92, generalized linear model (GLM) — To account for the non-normal distribution of the outcome, confidence intervals and p-values were obtained using a bias corrected and accelerated bootstrap resampling procedure with 10,000 replicates; generalized linear model (GLM) with an identity link; Maximum likelihood (MLE) = -0.035, 95% CI 2-sided [-0.727 to 0.657] — Confidence intervals and p-values were obtained using a bias-corrected and accelerated bootstrap resampling procedure with 10,000 replicates

2. Secondary Outcome: Treatment Satisfaction as Assessed by a Single Item From the International Outcome Inventory - Comprehensive Hearing Intervention (IOI-CHI) Scale
Description: The IOI-CHI is an interviewer-administered scale that consists of 6 items where participants self-report satisfaction with the hearing intervention using a 5-point Likert scale; treatment satisfaction is based on the item "Considering everything, do you think your present hearing intervention is worth the trouble?"), with scores ranging from 1 to 5 and higher scores indicating more treatment satisfaction.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Hearing Healthcare Group | Telehealth Hearing Healthcare Group
Number analyzed (Participants) | 159 | 153
score on a scale | 4.78 (0.47) | 4.78 (0.44)
Statistical Analysis 1: Comparison: Conventional Hearing Healthcare Group vs Telehealth Hearing Healthcare Group; Used a weighted regression model with an identity link to compare treatment satisfaction at one-year post-randomization between participants assigned to the telehealth HHC or conventional HHC. Inverse probability of treatment weights will be calculated and included in the model for the secondary outcome; Test type: Superiority; p = 0.87, generalized linear model (GLM); Maximum likelihood (MLE) = -0.011, 95% CI 2-sided [-0.147 to 0.125] — To account for the non-normal distribution of the outcome, confidence intervals and p-values were obtained using a bias corrected and accelerated bootstrap resampling procedure with 10,000 replicates

3. Secondary Outcome: Ability to Hear for Primary Communication Goal as Assessed by a Single Item From the Client-Oriented Scale of Improvement (COSI) Goals Achievement Questionnaire
Description: Achievement of COSI goals will be assessed by asking participants to rate their current ability to hear for their primary goal using a 5-point Likert scale, with options 1=hardly ever (10%), 2=occasionally (25%), 3=half of the time (50%), 4=most of the time (75%), and 5=almost always (95%), where higher scores indicate greater ability to hear. Mean of participant scale choice is reported.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Hearing Healthcare Group | Telehealth Hearing Healthcare Group
Number analyzed (Participants) | 159 | 153
score on a scale | 4.25 (0.74) | 4.29 (0.69)
Statistical Analysis 1: Comparison: Conventional Hearing Healthcare Group vs Telehealth Hearing Healthcare Group; Used a weighted regression model with an identity link to compare primary COSI goal achievement at one-year post-randomization between participants assigned to the telehealth HHC or conventional HHC. Inverse probability of treatment weights will be calculated and included in the model for the secondary outcome; Test type: Superiority; p = 0.66, generalized linear model (GLM); Maximum likelihood (MLE) = 0.059, 95% CI 2-sided [-0.201 to 0.320] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Hearing-specific Quality of Life as Assessed by the Hearing Handicap Inventory for the Elderly - Screening Version (HHIE-S) Questionnaire
Description: The HHIE-S is an interviewer-administered questionnaire that consists of 10 items; participants rate whether hearing loss affects them in different situations (yes, sometimes, or no); the total score is the sum of all responses and ranges from 0 to 40, with higher scores indicating greater hearing issues.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Hearing Healthcare Group | Telehealth Hearing Healthcare Group
Number analyzed (Participants) | 159 | 153
units on a scale | 7.33 (7.10) | 7.16 (6.49)
Statistical Analysis 1: Comparison: Conventional Hearing Healthcare Group vs Telehealth Hearing Healthcare Group; Used a weighted regression model with an identity link to compare hearing-specific quality of life at one-year post-randomization between participants assigned to the telehealth HHC or conventional HHC. Inverse probability of treatment weights will be calculated and included in the model for the secondary outcome; Test type: Superiority; p = 0.38, generalized linear model (GLM); Maximum likelihood (MLE) = -1.96, 95% CI 2-sided [-6.349 to 2.435] — [estimate comment as in outcome 2, analysis 1]

5. Other Pre Specified Outcome: Average Daily Hours of Hearing Aid Use Through Two Years of Follow-up
Description: as for outcome 1
Time Frame: Up to 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: Up to 1 year.
Description: Otitis externa and cerumen impaction or ear foreign body requiring removal by a physician were considered adverse events.
Arm/Group | Conventional Hearing Healthcare Group | Telehealth Hearing Healthcare Group
All-Cause Mortality (participants affected / at risk) | 0/176 | 4/163
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/163
Other Adverse Events (participants affected / at risk) | 7/176 | 11/163
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Hearing Healthcare Group (N=176) | Telehealth Hearing Healthcare Group (N=163)
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 2 (2) — An inflammation, irritation, or infection of the external ear canal
Cerumen impaction (Ear and labyrinth disorders) | 4 (4) | 7 (7) — Earwax blockage
Other (Ear and labyrinth disorders) | 2 (2) | 2 (2) — Type B tympanogram right ear requiring medical evaluation; Extremely low blood pressure; Abnormal tympanograms associated with recent illness; Myringotomy LEFT ear following sudden hearing loss

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT05070429/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT05070429/SAP_001.pdf